CLINICAL TRIAL: NCT04651790
Title: Multicenter, Phase 3, Randomized Clinical Study to Evaluate the Efficacy, Safety and Immunogenicity of Two Vaccination Schedules of an Inactivated Vaccine Against SARS-CoV-2 Infection in Adults.
Brief Title: Efficacy, Safety, and Immunogenicity of Two Vaccination Schedules of an Inactivated Vaccine Against COVID-19 in Adults
Acronym: CoronaVac3CL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Ministry of Health, Chile (Other Government); Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 200708006
Record Dates: First submitted 2020-11-20; First posted 2020-12-03 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2022-06

CONDITIONS: Covid19; Vaccines
Keywords: Clinical trials; Covid19; Inactivated vaccine
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaccine 0-14 (Active Comparator): Inactivated vaccine against SARS-CoV-2 2 doses on day 0 and 14
  Interventions: Biological: SARS-CoV-2 inactivated vaccine
- Vaccine 0-28 (Experimental): Inactivated vaccine against SARS-CoV-2 2 doses on day 0 and 28
  Interventions: Biological: SARS-CoV-2 inactivated vaccine

INTERVENTIONS:
Biological: SARS-CoV-2 inactivated vaccine — The vaccine contains inactivated SARS-CoV-2 virus, aluminum hydroxide, disodium hydrogen phosphate, sodium dihydrogen phosphate and sodium chloride.The final product will be supplied in a pre-filled syringe containing 0.5 ml of solution for injection that corresponds to a dose of the vaccine.
  Other Names: Coronavac

SUMMARY:
The study will evaluate the efficacy, safety, and immunogenicity of two vaccination schedules of an inactivated vaccine against SARS-CoV-2 infection in adults. Two doses of the vaccine will be administered in a 0,14 and a 0,28-day schedule. Follow-up of safety and efficacy will be assessed for 12 months after the first dose. Immunogenicity will be studied in a subgroup of participants.

DETAILED DESCRIPTION:
This study will evaluate the efficacy, safety, and immunogenicity of two vaccination schedules of an inactivated vaccine against SARS-CoV-2 infection in adults. This study will be performed in 8 centers. Two schedules will be compared: 0,14 and 0,28-day, at a 1:1 rate. 40% of participants will be 60 or more years-old. Follow-up of safety and efficacy will be assessed for 12 months after administering the first dose. The collection of the data will be through an electronic Case Report Form. Immunogenicity will be studied in a subgroup of participants. Initially, 2,300 volunteers will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age.
* Demonstrate the capacity to understand and sign the Informed Consent document.
* Agree to comply with the study procedures and visits.

Exclusion Criteria:

* History of confirmed symptomatic SARS CoV-2 infection.
* Pregnant (confirmed by positive urine pregnancy test) or breastfeeding females, and/or expressing intention to have sexual practices with reproductive potential without using contraceptive methods in the three months following vaccination.
* History of an allergic reaction to the vaccine or components of the study vaccine or placebo.
* Evidence of uncontrolled neurological, cardiac, pulmonary, hepatic, or renal disease, according to anamnesis or physical examination; Significant changes in treatment or hospitalizations due to worsening of the condition in the last three months are indicators of uncontrolled disease.
* Diseases that impair the immune system including neoplasms (except basal cell carcinoma), congenital or acquired immunodeficiencies, and uncontrolled autoimmune diseases not controlled according to anamnesis or physical examination.
* Behavioral, cognitive, or psychiatric illness that, in the opinion of the principal investigator or his medical representative, affects the participant's ability to understand and collaborate with the requirements of the study protocol.
* Use of immunosuppressive therapies six months before inclusion in the study or its scheduled use within two years of inclusion. Immunosuppressive therapies will be considered: antineoplastic chemotherapy, radiation therapy, immunosuppressants to induce tolerance to transplants, among others.
* Have received an immunosuppressive dose of corticosteroids in the last three months before inclusion in the study or scheduled administration of an immunosuppressive dose of corticosteroids for the three months following inclusion in the study. The dose of corticosteroids considered immunosuppressive is equivalent to prednisone at a dose of 20 mg/day for adults for more than a week. The continuous use of topical or nasal corticosteroids is not considered immunosuppressive.
* History of asplenia, either anatomic or functional.
* History of bleeding disorders, as deficiency of clotting factors, coagulopathy, platelet dysfunction, or previous history of bleeding or significant bruising after IM injection or venipuncture.
* Any alcohol or drug abuse in the last 12 months before inclusion in the study that has caused medical, professional, or family problems, as indicated by clinical history.
* Have received blood products (transfusions or immunoglobulins) in the last three months before inclusion in the study.
* Have received any vaccine with a live attenuated virus in the last 28 days or inactivated vaccine in the last 14 days before their inclusion in the study, or have immunization scheduled for the first 28 days after their inclusion in the study.
* Participation in another clinical trial with product administration under investigation during the six months before its inclusion in the study or scheduled participation in another clinical trial in the two years following inclusion.
* Previous participation in a COVID-19 vaccine evaluation study or previous exposure to a COVID-19 vaccine.
* Fever (>37.8°C) within 72 hours before vaccination.
* Any other condition that, in the opinion of the principal investigator or his medical representative, could jeopardize the safety or rights of a potential participant or that would prevent him from complying with this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2300 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Frequency of solicited and unsolicited adverse events that occur during the period of one week after each dose of the vaccine in two vaccination schedules: 0,14 and 0,28 days stratified by age group (18-59 years, and 60 or more years). | During the first 7 days after each dose of vaccine
  The frequency of solicited and unsolicited local and systemic adverse reactions will be registered. This will be measured during the first 7 days after each vaccination. These adverse reactions will be registered according to the age group in adults (18-59 years old) and the elderly (60 years of age or older).
Incidence of symptomatic cases of virologically confirmed COVID-19 two weeks after the second dose of each vaccination schedule. | Two weeks after second dose up to one year after first dose
  Vaccine efficacy to prevent virologically confirmed COVID-19 two weeks after the second dose of each vaccination schedule will be determined

SECONDARY OUTCOMES:
Incidence of hospitalized cases of COVID-19 two weeks after the second vaccination of two vaccination schedules | Since two weeks after the second dose of two vaccination schedules and up 12 month after first dose
  The incidence of hospitalized cases of COVID-19 two weeks after the second vaccination of two vaccination schedules will be determined.
Incidence of severe cases or deaths of COVID-19 virologically confirmed two weeks after the second vaccination of two vaccination schedules | Since two weeks after the second dose up 12 month after first dose
  The incidence of severe cases of COVID-19 and deaths, confirmed through PCR, two weeks after the second vaccination of two vaccination schedules, will be determined.
Incidence of adverse reactions to the vaccine, local and systemic, solicited and unsolicited, within the period of four weeks after each vaccination of two vaccination schedules, according to the age, adults (18-59 years old) and elder (>60 years) | Four weeks after each dose of vaccine in two vaccination schedules
  The incidence of adverse reactions to the vaccine, both local and systemic, solicited and unsolicited will be determined. These adverse reactions will be measured within the period of four weeks after each dose of vaccination of two vaccination schedules. These adverse reactions will be registered according to the age group in adult (18-59 years old) and elder (60 years of age or older) subjects
Frequency of severe COVID-19 cases in participants who received at least one dose of vaccine in two vaccination schedules | Since first dose up to 12 month after
  The frequency of severe COVID-19 cases in participants who received at least one dose of vaccine in two vaccination schedules will be determined.
Incidence of serious adverse events (SAE) and adverse events in participants who have received at least one dose of the vaccine, in two vaccination schedules | Since first dose up to 12 month after
  The occurrence of serious adverse events (SAE) and adverse events of special interest in participants who have received at least one dose of the vaccine in two vaccination schedules, will be determined
Percentage of participants that show a significant increase in SARS-CoV-2 specific T cells after vaccination, in two vaccination schedules, determined by flow Cytometry and ELISPOT | Since first dose up to 4 weeks after second dose
  The cellular immune response in a subgroup of participants, before and two and four weeks after the administration of each dose of the vaccine, in two vaccination schedules will be evaluated
Percentage of participants with a significant increase of anti-SARS-CoV-2 antibodies, determined by ELISA | Since first dose up to 2 weeks after second dose
  The presence of anti-SARS-CoV-2 antibodies in a subgroup of participants, before and two weeks after the administration of each dose of the vaccine, in two vaccination schedules, will be evaluated.
Percentage of participants that show a significant increase in SARS-CoV-2 specific T cells after vaccination, determined by flow Cytometry and ELISPOT | Since first dose up to 4 weeks after second dose
  The cellular immune response in a subgroup of participants, before and two and four weeks after the administration of each dose of the vaccine, will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Katia Abarca, MD, Study Director — Pontificia Universidad Catolica de Chile; Alexis M Kalergis, PhD, Study Director — Pontificia Universidad Catolica de Chile; Susan M Bueno, PhD, Study Director — Pontificia Universidad Catolica de Chile; Pablo A González, PhD, Study Director — Pontificia Universidad Catolica de Chile
Locations (1):
- Centro de Especialidades Médicas, Red de Salud UC Christus, Santiago, RM, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Galvez NMS, Pacheco GA, Schultz BM, Melo-Gonzalez F, Soto JA, Duarte LF, Gonzalez LA, Rivera-Perez D, Rios M, Berrios RV, Vazquez Y, Moreno-Tapia D, Vallejos OP, Andrade CA, Hoppe-Elsholz G, Iturriaga C, Urzua M, Navarrete MS, Rojas A, Fasce R, Fernandez J, Mora J, Ramirez E, Gaete-Argel A, Acevedo ML, Valiente-Echeverria F, Soto-Rifo R, Weiskopf D, Grifoni A, Sette A, Zeng G, Meng W; CoronaVacCL03 Study Group; Gonzalez-Aramundiz JV, Johnson M, Goldblatt D, Gonzalez PA, Abarca K, Bueno SM, Kalergis AM. Differences in the immune response elicited by two immunization schedules with an inactivated SARS-CoV-2 vaccine in a randomized phase 3 clinical trial. Elife. 2022 Oct 13;11:e81477. doi: 10.7554/eLife.81477. PMID 36226829
- [Derived] Luan N, Li T, Wang Y, Cao H, Yin X, Lin K, Liu C. Th2-Oriented Immune Serum After SARS-CoV-2 Vaccination Does Not Enhance Infection In Vitro. Front Immunol. 2022 Apr 8;13:882856. doi: 10.3389/fimmu.2022.882856. eCollection 2022. PMID 35464483
- [Derived] Bueno SM, Abarca K, Gonzalez PA, Galvez NM, Soto JA, Duarte LF, Schultz BM, Pacheco GA, Gonzalez LA, Vazquez Y, Rios M, Melo-Gonzalez F, Rivera-Perez D, Iturriaga C, Urzua M, Dominguez A, Andrade CA, Berrios RV, Canedo-Marroquin G, Covian C, Moreno-Tapia D, Saavedra F, Vallejos OP, Donato P, Espinoza P, Fuentes D, Gonzalez M, Guzman P, Munoz-Venturelli P, Perez CM, Potin M, Rojas A, Fasce R, Fernandez J, Mora J, Ramirez E, Gaete-Argel A, Oyarzun-Arrau A, Valiente-Echeverria F, Soto-Rifo R, Weiskopf D, Sette A, Zeng G, Meng W, Gonzalez-Aramundiz JV, Kalergis AM. Interim report: Safety and immunogenicity of an inactivated vaccine against SARS-CoV-2 in healthy chilean adults in a phase 3 clinical trial. medRxiv [Preprint]. 2021 Apr 1:2021.03.31.21254494. doi: 10.1101/2021.03.31.21254494. PMID 35441164
- [Derived] Duarte LF, Galvez NMS, Iturriaga C, Melo-Gonzalez F, Soto JA, Schultz BM, Urzua M, Gonzalez LA, Vazquez Y, Rios M, Berrios-Rojas RV, Rivera-Perez D, Moreno-Tapia D, Pacheco GA, Vallejos OP, Hoppe-Elsholz G, Navarrete MS, Rojas A, Fasce RA, Fernandez J, Mora J, Ramirez E, Zeng G, Meng W, Gonzalez-Aramundiz JV, Gonzalez PA, Abarca K, Bueno SM, Kalergis AM. Immune Profile and Clinical Outcome of Breakthrough Cases After Vaccination With an Inactivated SARS-CoV-2 Vaccine. Front Immunol. 2021 Sep 29;12:742914. doi: 10.3389/fimmu.2021.742914. eCollection 2021. PMID 34659237